CLINICAL TRIAL: NCT06085053
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics of TQA3038 Injection in Healthy Adult Subjects.
Brief Title: A Clinical Trial of TQA3038 Injection in Healthy Adult Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQA3038-I-01
Record Dates: First submitted 2023-10-11; First posted 2023-10-16 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-10

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQA3038 injection (Experimental): One dose of TQA3038 injection in Day 1.
  Interventions: Drug: TQA3038 injection
- TQA3038 injection matching placebo (Placebo Comparator): One dose of TQA3038 injection matching placebo in Day 1.
  Interventions: Drug: TQA3038 injection matching placebo

INTERVENTIONS:
Drug: TQA3038 injection — TQA3038 is an injection.
  Arms: TQA3038 injection
Drug: TQA3038 injection matching placebo — Placebo injection contains no active substance.
  Arms: TQA3038 injection matching placebo

SUMMARY:
This is a phase 1 study in which healthy adult subjects will receive TQA3038 or placebo and will be assessed for safety, tolerability, pharmacokinetics.

In the single ascending dose (SAD) part, healthy adult subjects will receive one dose of TQA3038 or placebo, administered subcutaneously (SC).

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18～60 years.
* Body mass index (BMI) 19 - 26 kg/m^2.

Exclusion Criteria:

* Any clinically significant chronic or acute medical condition that makes the volunteer unsuitable for participation；
* History or evidence of drug or alcohol abuse；
* History of intolerance to SC injection；

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Up to 85 days.
  Number of subjects with adverse events (AEs) and serious adverse events (SAEs) assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Number of subjects with clinically significant abnormalities | Up to 85 days.
  Number of subjects with clinically significant abnormalities in vital signs, electrocardiogram (ECG), and laboratory parameters graded by CTCAE v5.0.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Predose on Day 1 and 30 minutes, 1, 2, 4, 6, 8, 10, 12, 24, 48 hours postdose
  Maximum concentration of TQA3038 and its metabolite in plasma
Time to Reach Maximum Plasma Concentration (Tmax) | Predose on Day 1 and 30 minutes, 1, 2, 4, 6, 8, 10, 12, 24, 48 hours postdose
  Time to reach Cmax of TQA3038 and its metabolite in plasma
Area Under the Plasma Concentration Versus Time Curve (AUC) | Predose on Day 1 and 30 minutes, 1, 2, 4, 6, 8, 10, 12, 24, 48 hours postdose
  Area under the curve of TQA3038 and its metabolite from time 0 to last measurable time
Apparent Terminal Elimination Half-life (T1/2) | Predose on Day 1 and 30 minutes, 1, 2, 4, 6, 8, 10, 12, 24, 48 hours postdose
  Apparent Elimination Half-life (T1/2) of TQA3038 in Plasma
Apparent Plasma Clearance (CL/F) | Predose on Day 1 and 30 minutes, 1, 2, 4, 6, 8, 10, 12, 24, 48 hours postdose
  Apparent Plasma Clearance (CL/F) of TQA3038 in Plasma
Fraction eliminated in the urine | Predose, 0-4 hours, 4-8 hours, 8-12 hours, 12-24 hours, 48 hours and 168 hours after dose on Day 1.
  Apparent Plasma Clearance (CL/F) of TQA3038 in Plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China